CLINICAL TRIAL: NCT05165875
Title: Splint Versus Steroid Injection for DeQuervain's Tenosynovitis: A Randomized Trial
Brief Title: Splint Versus Steroid Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/00246
Record Dates: First submitted 2021-12-01; First posted 2021-12-21 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2021-12

CONDITIONS: De Quervain Syndrome
MeSH Terms: interventions — Splints

STUDY DESIGN:
Intervention Model Description: The trial design is a multicentre, randomized controlled, assessor blinded, 2 arm 1:1 superiority trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized: Steroid injection (Other): 1ml injection of a mixture of 0.5ml triamcinolone acetonide (50mg/5ml) and 0.5ml 1% lignoacaine is given intra-thecally into the first extensor compartment.
  Interventions: Drug: Hydrocortisone-Lidocaine
- Randomized: Splint (Other): a long thumb spica thermoplastic splint (wrist neutral, 30º CMCJ flexion, 30º thumb abduction, IPJ free) will be customized and intermittent active range of motion exercises will be taught for 4 weeks
  Interventions: Other: Splint

INTERVENTIONS:
Drug: Hydrocortisone-Lidocaine — Intervention will be done on the same day based on the randomization.
  For the steroid injection group, a 1ml injection of a mixture of 0.5ml triamcinolone acetonide (50mg/5ml) and 0.5ml 1% lignoacaine is given intra-thecally into the first extensor compartment.
  For both groups, routine analgesia is not prescribed but the use is not restricted to the participants.
  Arms: Randomized: Steroid injection
Other: Splint — Intervention will be done on the same day based on the randomization. For the splint group, a long thumb spica thermoplastic splint (wrist neutral, 30º CMCJ flexion, 30º thumb abduction, IPJ free) will be customized and intermittent active range of motion exercises will be taught for 4 weeks. Subsequently, the splint will be weaned and passive range of motion exercises taught.
  For both groups, routine analgesia is not prescribed but the use is not restricted to the participants.
  Arms: Randomized: Splint

SUMMARY:
The primary aim is to compare the effectiveness of splinting versus steroid injection in improving the DASH scores in participants diagnosed with De Quervain's tenosynovitis over a period of 6 months.

DETAILED DESCRIPTION:
The primary hypothesis is that steroid injection into the first dorsal compartment is more effective compared with splinting at 3 months.

The secondary hypothesis is that steroid injection yields better clinical outcomes compared with splinting at 1 month, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of de Quervain's tenosynovitis based on the de Quervain's screening tool (DQST) with scores ≥ 5 (refer to table 1)
* No prior treatment
* Above 21 years of age

Exclusion Criteria:

* Allergy to steroid (triamcinolone acetate) or local anaesthetic (lignocaine)
* History of work related trauma

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Quick Disability of Arm, Shoulder, Hand (QuickDASH) | 6 months
  Our co- primary outcome would be QuickDash. QuickDash is a disability score we use for the upper limb where the higher score indicates greater disability and severity. We would expect a decrease in QuickDash scores following a success in the treatment measure. The resultant score is reported on a scale of 0 to 100, where 0 represents no disability and 100 represents total disability
Patients who have recovered from De Quervain's Tenosynovitis | 6 months
  The other primary outcomes would be the number of patients who have completely recovered from De Quervain's tenosynovitis. This will be determined by the global improvement the patient feels that will be ranked on a 7 point Likert scale (1: very much worse, 2: much worse, 3:slightly worse, 4:no change, 5:slightly better, 6:much better, 7:completely resolved).

CONTACTS AND LOCATIONS:
Overall Officials: Renita Sirisena, Principal Investigator — National University Hospital, Singapore